CLINICAL TRIAL: NCT03977844
Title: Community Resilience Learning Collaborative and Research Network
Acronym: C-LEARN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: National Academies of Sciences - Gulf Research Program (Unknown); University of California, Los Angeles (Other); University of Southern California (Other)
Responsible Party: Principal Investigator, Benjamin Springgate, Associate Professor, Louisiana State University Health Sciences Center in New Orleans
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2000008324
Record Dates: First submitted 2019-05-30; First posted 2019-06-06 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Depression; Social Stress; Anxiety; Quality of Life; Disaster
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Health Planning Technical Assistance; Community Resources

STUDY DESIGN:
Intervention Model Description: Community agencies are randomized to participate in either of two intervention arms. Clients recruited at agencies in either community-level intervention arm are randomized at individual level to participate in one of two technology interventions. 2 arms at community level of randomization, 2 arms at individual level of randomization.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Client-level participants are unaware of which arm to which the agencies from which they have been recruited have been assigned at the community agency level randomization.
  Providers are unaware of which clients have been recruited into the study, as well as to which arm the clients have been assigned at the individual level randomization for the technological mobile phone intervention.
  Outcomes assessors at follow-up assessments are unaware of which arm the participants have been assigned at either the community or individual level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Technical Assistance (Active Comparator): Technical Assistance. At the community program level of randomization, community agencies and their staff will be invited to access weekly webinars and toolkits to improve their abilities to support clients' depression care, disaster preparedness and recovery, financial security, and housing security.
  Interventions: Other: Technical Assistance
- Community Engagement and Planning (Experimental): Community Engagement and Planning. At the community program level of randomization, community agencies and their staff will be invited to access weekly webinars and toolkits to improve their abilities to support clients' depression care, disaster preparedness and recovery, financial security, and housing security. In addition, community agencies will be invited to meet with one another to develop novel and investigator supported coalitions using principles of community partnered participatory research that will adapt toolkits and other local assets to seek to enhance community resilience related to threats of disaster risk, financial insecurity, housing insecurity, mental health, or other coalition-determined domains.
  Interventions: Other: Technical Assistance; Other: Community Engagement and Planning
- Community Resources (CR) (Active Comparator): Community Resources (CR). At the Individual level of randomization, individuals in the Community Resources (CR) arm will receive access to toolkits and local resources related to depression care, disaster preparedness and recovery, financial security, and housing security.
  Interventions: Other: Community Resources (CR)
- Community Resources (CR) + eBT (Experimental): Community Resources + eBT. At the Individual level of randomization, individuals in the CR+eBT arm will receive access to toolkits and local resources related to depression care, disaster preparedness and recovery, financial security, and housing security, along with an interactive component to support CBT-informed coping with mood and stressors at the individual level.
  Interventions: Other: Community Resources (CR); Other: Community Resources + eBT

INTERVENTIONS:
Other: Technical Assistance — TA for Individual Programs TA uses experts to train program staff via webinars and site visits, using the same toolkits as CEP, in a "train the trainer" approach. TA provides a series of webinars and as needed site visits, focused in the example of depression care on team support for assessment, treatment support as appropriate with medication and/or psychotherapy, case management and educational resources and access to intervention toolkits. It also includes webinars and training toolkits for agencies on domains of social risk factors for health (financial security and housing security) as well as disaster preparedness and recovery.
  Arms: Community Engagement and Planning; Technical Assistance
Other: Community Engagement and Planning — CEP for Coalitions CEP creates multi-sector networks to collaborate in evidence-based and community-prioritized toolkits or intervention materials. CEP supports a series of biweekly to monthly meetings to develop network and individual program capacity, prepare stakeholders as co-leads, and create a written training plan following CPPR principles [48, 64]. CEP councils consider local context, i.e., cultural assets and stakeholder input. Disaster preparedness and public health sectors will be encouraged to offer education/resources on social determinants and disasters within CEP training plans. CEP will be supported by a Learning Collaborative, meeting 2-3 times, using activities such as project examples, tabletop exercises and self-assessment to identify gaps and formulate goals for improvement.
  Arms: Community Engagement and Planning
Other: Community Resources (CR) — The CR app will primarily provide informational resources and referral information relevant to the local community. We will identify resources for depression, social determinants and disaster preparedness and response within each community during planning with local stakeholders.
  Arms: Community Resources (CR); Community Resources (CR) + eBT
Other: Community Resources + eBT — The CR+eCBT app consists of the functionality of the CR app along with an interactive component to support CBT-informed coping with mood and stressors at the individual level. This component was developed previously by our group using participatory methods with community partners and includes interactive support to enhance social support networks, support cognitive restructuring (framed through partnered input as "Catch it, Check it, Change it"), and encourage pleasant activities [65]. Participants will receive text message notifications (with frequency set by participants, up to several times per day) and can either reply back to messages to explore content or click a link in the message to access the interactive mobile app.
  Arms: Community Resources (CR) + eBT

SUMMARY:
C-LEARN is designed to determine how to build service program and individual client capacity to improve mental health-related quality of life among individuals at risk for depression, with exposure to social risk factors or concerns about environmental hazards in areas of Southern Louisiana at risk for events such as hurricanes and storms. The study uses a Community Partnered Participatory Research (CPPR) framework to incorporate community priorities into study design and implementation. The first phase of C-LEARN is assessment of community priorities, assets, and opportunities for building resilience through key informant interviews and community agency outreach. Findings from this phase will inform the implementation of a two-level (program-level and individual client level) randomized study in up to six South Louisiana communities. Within communities, health and social-community service programs will be randomized to Community Engagement and Planning (CEP) for multi-sector coalition support or Technical Assistance (TA) for individual program support to implement evidence-based and community-prioritized intervention toolkits, including an expanded version of depression collaborative care and resources (referrals, manuals) to address social risk factors such as financial or housing instability and for a community resilience approach to disaster preparedness and response. Within each arm, the study will randomize individual adult clients to one of two mobile applications that provide informational resources on services for depression, social risk factors, and disaster response or also provide psychoeducation on Cognitive Behavioral Therapy to enhance coping with stress and mood. Planned data collection includes baseline, 6-month and brief monthly surveys for clients, and baseline and 12-month surveys for administrators and staff. Due to COVID-19 pandemic interruption of the study, the recruitment into the randomized controlled trials was halted. A third study part was added to assess the impact of the pandemic on participating study agencies and the community.

DETAILED DESCRIPTION:
C-LEARN's overall aim is to determine how best to improve resilience, particularly mental health-related quality of life for individual adult clients of diverse health and community-social service programs, through alternative strategies to build capacity of programs to provide services for depression, social risk factors and disaster-related concerns, as well as through alternative forms of individual client information technology support for addressing the same range of issues.

Specific aims are:

To engage communities in South Louisiana in a community learning initiative on how to best build capacity to enhance resilience to depression, adverse social determinants of health, and disaster exposure. This aim includes a qualitative assessment of local community resilience priorities and assets to inform study implementation.

To compare the effectiveness for improving mental health quality of life (MHRQL) (primary) and coping with stressors and other resilience outcomes (secondary), of two program-level interventions to build capacity for resilience programs: 1) Technical Assistance (TA) to individual programs vs 2) Community Engagement and Planning (CEP) to support multi-sector coalitions.

To compare the effectiveness for improving MHRQL and other resilience outcomes of two mobile apps: CR and CR+eCBT: 1) CR - An app providing only information on community resources, or 2) CR+eCBT - An app providing information on community resources and education on a cognitive behavioral therapy (eCBT) based approach to enhance individual resilience (i.e., coping with mood and stressors).

To describe strategies CEP coalitions used to address depression, social determinants and disaster resilience, to inform interpretation and dissemination of findings.

Design

The design has an overall CPPR approach to implement a 2 by 2, randomized comparative effectiveness trial. Randomization occurs at the program level to either CEP or TA, where a program is a discrete services program with its own staff and clients; there may be multiple programs within a given administrative agency, including different geographic sites such as clinics. Further, programs may offer services in different content areas, such as physical health, mental health, social services, disaster services, faith-based, etc., referred to as different "sectors." In addition, individual participants will be randomized to one of two mobile apps for coping with stressors and disasters.

The project and design phase has been led by a Leadership Council, including academic, community, and health system participants who have guided all aspects of the study, and operate under CPPR principles.1 Initial leaders are academic and community partners from the Community and Patient Partnered Research Network (CPPRN) across South Louisiana and Los Angeles with additional stakeholder advisors from New Orleans, Baton Rouge and Coastal South Louisiana planned for as engagement of communities proceeds.2 The Council reviews work group recommendations and facilitates larger community input and approval through a stakeholder advisory committee and larger community conferences, one of which occurred prior to publishing this phase (pre-program recruitment) of the protocol.

Interventions

The main comparators are CEP and TA. Healthcare and community-based programs that are assigned to CEP and TA will both receive training and support for implementation of an expanded model of evidence-based depression collaborative care that also addresses social determinants and disaster readiness. The depression toolkits to be used are from studies on adults, including, racial/ethnic minority and low-income groups, with community health worker manuals from prior work in New Orleans, adapted for community-based programs in the Community Partners In Care (CPIC) study.3-7 Toolkits use a team-based, stepped-care approach supporting assessment, referral and treatment, outcomes monitoring and care adjustment with specialty supervision and case managers for coordination and client education. While based on components of collaborative care for depression (clinical assessment and medication management for physicians; clinical assessment and CBT for licensed counselors; case management support for screening, education and patient activation, problem solving, care coordination and outreach; team management support), the interventions will also include resources to address main social determinants (e.g., poverty/financial planning, housing resources) and disaster preparedness/response, such as online resources developed after LACCDR.8 Initial adaptations have been made with stakeholder input, but work groups will continue to refine some materials prior to client recruitment. The differences between CEP and TA are described in the following sections.

CEP for Coalitions CEP creates multi-sector networks to collaborate in evidence-based and community-prioritized toolkits or intervention materials.9,10 CEP supports a series of biweekly to monthly meetings to develop network and individual program capacity, prepare stakeholders as co-leads, and create a written training plan following CPPR principles.1,11 CEP councils consider local context, i.e., cultural assets and stakeholder input. Disaster preparedness and public health sectors will be encouraged to offer education/resources on social determinants and disasters within CEP training plans. CEP will be supported by a Learning Collaborative, meeting 2-3 times, using activities such as project examples, tabletop exercises and self-assessment to identify gaps and formulate goals for improvement. 8,11

TA for Individual Programs TA uses experts to train program staff via webinars and site visits, using the same toolkits as CEP, in a "train the trainer" approach with outside referral for intensive support such as for full supervision in CBT. TA provides a series of webinars and as needed primary care site visits, focused on team support for assessment, treatment support as appropriate with medication and/or psychotherapy, case management and educational resources and access to intervention toolkits. TA experts may include a psychiatrist, CBT expert therapist, case manager, support staff and community leader to engage service programs. The team will include experts on components such as financial planning and disaster preparedness.

Individual-Level Mobile Apps

C-LEARN will compare two mobile apps created as part of this study (referred to as CR and CR+eCBT) that permit interactive text messaging, mobile web, or interactive voice response (IVR) interactions, using an information technology platform (Chorus) specifically designed for participatory development.2 Each mobile app will be adapted through workgroups with stakeholders in order to tailor content to each community. The CR app will primarily provide informational resources and referral information relevant to the local community. The study team and investigators will identify resources for depression, social determinants and disaster preparedness and response within each community during planning with local stakeholders. The CR+eCBT app consists of the functionality of the CR app along with an interactive component to support CBT-informed coping with mood and stressors at the individual level. This component was developed previously by our group using participatory methods with community partners and includes interactive support to enhance social support networks, support cognitive restructuring (framed through partnered input as "Catch it, Check it, Change it"), and encourage pleasant activities 12. Participants will receive text message notifications (with frequency set by participants, up to several times per day) and can either reply back to messages to explore content or click a link in the message to access the interactive mobile app.

Measures and outcomes (primary/secondary) are identified elsewhere in the clinicaltrials.gov submission. Randomization, sampling, and proposed statistical analysis details are available in the protocol, also included with this submission.

Part three added during the pandemic consisted of qualitative interviews to assess the impact of the pandemic on organizations and communities in Southeast Louisiana.

Human Subjects Protection All procedures will have prior review and approval from the LSU Health Sciences Center-New Orleans (LSUHSC-NO) Institutional Review Board (IRB), and partnering research institutions will enter into reliance agreements with LSUHSC-NO. The study currently has IRB approval to conduct qualitative interviews, and to consent and enroll participating agencies, administrators, and providers.

ELIGIBILITY:
Inclusion Criteria - Providers or Administrators:

* 18 years of age or older
* English reading and writing fluency
* Resident of Southeast Louisiana
* Employed at a participating community agency

Inclusion Criteria - Clients:

* 18 years of age or older
* English fluency in reading and writing
* Resident of Southeast Louisiana
* Client of a participating community agency
* Access to a phone that receives SMS text messages
* (PHQ-8 ≥ 10 OR MCS-12 ≤ 40) OR
* (Disaster exposure AND housing insecurity) OR
* (Disaster exposure AND financial insecurity)

Exclusion Criteria - All:

* Does not meet inclusion criteria above
* Grossly intoxicated
* Mentally incapacitated

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Mental Health Related Quality of Life | Baseline and 6 months.
  Changes in mental health-related quality of life defined by Short Form Survey (SF-12), Mental Health Composite Score (MCS). Survey scored from 0-100 using algorithm for comparison to normative data. Scores interpreted in relation to the normative mean score of 50. >50 = better mental health quality of life than the mean; <50 indicates worse physical or mental health quality of life than the mean.
Depression | Baseline and 6 months.
  Depression severity defined by the Personal Health Questionnaire-8 (PHQ-8). Each item is scored 0-3 (0= not at all; 3= nearly every day), yielding a possible total between 0 and 24. PHQ-8 score of 10 or greater indicates at least moderate depression. Score of 20 or more indicates likely severe or major depression.

SECONDARY OUTCOMES:
Resilience | Baseline and 6 months.
  Individual resilience measured using the Brief Resilience Scale (BRS) on a 1-5 point scale. Scores below 3 indicate low resilience; scores above 4.3 indicate high resilience.
Physical Health Related Quality of life | Baseline to 6 months.
  Physical health-related quality of life defined by Short Form Survey (SF-12), Physical Health Composite Score (PCS). Survey scored from 0-100 using an algorithm for comparison to normative data. Scores are interpreted in relation to the normative mean score of 50. >50 = better physical health quality of life than the mean; <50 indicates worse physical or physical health quality of life than the mean.
Mental Wellness Indicator | Baseline and 6 months.
  Self-reported indicator of mental wellness; a response of at least "sometimes in the prior 4 weeks" on feeling calm or peaceful, having energy, or being happy.
Social Determinants of Health | Baseline and 6 months.
  Self-reported social factors that potentially affect health outcomes (mental and physical), access to care, accuracy of care, quality of care. Determined by self-report in screening survey, baseline and followup measures.
Behavioral Health Hospitalization | Baseline and 6 months.
  Avoiding any behavioral health hospitalization, with a sensitivity analysis of avoiding having ≥ four hospital nights.
Work loss days | Baseline and 6 months.
  For those employed, number of work-loss days in the prior 30 days.
General Anxiety Disorder (GAD-2) | Baseline and 6 months.
  General anxiety disorder is measured using the Generalized Anxiety Disorder (GAD-2). Each item is scored 0-3 yielding a possible total between 0 and 6. Scores 0-3 indicate low probability of anxiety disorder. Scores 3-6 indicate probable anxiety disorder.
Post Traumatic Stress Disorder | Baseline and 6 months.
  Post Traumatic Stress Disorder (PTSD) measured using Primary Care - Post Traumatic Stress Disorder Screen (PC-PTSD-5) screen for PTSD in a primary care setting. Items are scored 0 or 1 ("no" or "yes", respectively) yielding a potential total score of 5. Score of less than 3 indicates low probability of PTSD. Score of 3 or more indicates possible PTSD.
Body Mass Index | Baseline and 6 months.
  Body Mass Index (BMI) measured using Weight (in pounds) and height (in feet and inches) are self-reported by participant. Weight and height will be combined to report BMI in kg/m^2. Scores are considered on a continuous scale; scores under 18.5 are classified as underweight, scores 18.5-25 are classified as normal, scores 25-30 are considered overweight; > 30 is classified as obese.
Cigarette Smoking- Short Term | Baseline and 6 months.
  Self-reported number of cigarettes per day in the last 7 days.
Cigarette Smoking- Lifetime | Baseline and 6 months.
  Self-reported smoking of 100 cigarettes or more in lifetime. Scored 1 or 0; "yes" or "no" respectively.
Physical Activity | Baseline and 6 months.
  Self-reported regular activity level. Scored from 1 (not active at all) to 6 (extremely active).
Perceived Community Resilience Capacity | Baseline and 6 months.
  Perception of community capacity for resilience adapted from Communities Advancing Resilience Toolkit (CART). Each item scored 1 to 4; 1=strongly agree 4=strongly disagree yielding total score 0 to 20. Lower score indicates more favorable perception of community resilience capacity.
Self-efficacy | Baseline and 6 months.
  Self-efficacy in coping with depression social risk factors and disaster threats. Self-reported confidence in ability (self-efficacy) to overcome or control depression, take effective action to treat depression, and manage side-effects of antidepressant medication(s). Scored from 1 to 4, 1= Not at all confident, 4 = extremely confident. Three items averaged; higher mean indicates greater self-efficacy.
Coping | Baseline and 6 months.
  Self-report of individual coping skills used and response to stressful situations using a Likert scale scored 1-5, 1= never, 5= very often. Five items averaged; higher mean indicates more frequent use of coping skills.
Service use | Baseline and 6 months.
  Self-reported frequency of use and care satisfaction with health and social-community, housing, financial, and disaster services.
Life difficulties | Baseline and 6 months.
  Self-report of life difficulties in the previous 6 months. Includes exposure to disasters, violence, child custody changes, death, employment loss. Scored 1 or 0; "yes" or "no" respectively. Five items averaged; higher mean indicates more life difficulties.

OTHER OUTCOMES:
Medication for a mental health disorder | Baseline and 6 months.
  Self-reported use or prescription of any antidepressant, mood stabilizer, and any antipsychotic in the previous 6 months.
Barriers to care | Baseline and 6 months.
  Self-report of potential barriers to pursuing or receiving care, quality of care, or delayed service provision.
Alcohol use | Baseline and 6 months.
  Occurrence and severity of alcohol use adapted from the Alcohol Use Disorders Identification Test (AUDIT). Self-report of number of drinks consumed on a typical day, and frequency of alcohol use within a week or month. Latter two items scored 0 to 4, 0 = never 4=daily or almost daily/4 or more times a week. Total possible score = 0 to 8. Score of 3 AND >5 drinks per day = heavy or hazardous drinking.
Substance use | Baseline and 6 months.
  Occurrence or severity of potential substance use and substance use disorder measured using Drug Screening Questionnaire (DAST). Scored 1 or 0; "yes" or "no" respectively; total score 0-10. 0=low risk; 1-2 = risky; 3-5 = harmful; 6-10 = severe.
Social Support | Baseline and 6 months.
  Individual perceived social support measure adapted from Medical Outcomes Study (MOS) Social Support Survey. Scored 1-6; 1= all of the time, 6= none of the time. Average of all scores collected. Lower average indicates higher perceived social support.
Chronic health conditions | Baseline and 6 months.
  Self-report of a series of chronic health conditions including but not limited to diabetes, hypertension, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Springgate, MD, Principal Investigator — LSUHSC
Locations (1):
- Lsuhsc-No, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Springgate BF, Arevian AC, Wennerstrom A, Johnson AJ, Eisenman DP, Sugarman OK, Haywood CG, Trapido EJ, Sherbourne CD, Everett A, McCreary M, Meyers D, Kataoka S, Tang L, Sato J, Wells KB. Community Resilience Learning Collaborative and Research Network (C-LEARN): Study Protocol with Participatory Planning for a Randomized, Comparative Effectiveness Trial. Int J Environ Res Public Health. 2018 Aug 7;15(8):1683. doi: 10.3390/ijerph15081683. PMID 30720791
- [Background] Acosta JD, Augustine LA, Birch TL, et al. Strengthening the Response to Disasters and Trauma. In: Plough AL, ed. Community Resilience. Oxford University Press; 2021:140-153. doi:10.1093/oso/9780197559383.003.0012
- [Result] Palinkas LA, Springgate BF, Sugarman OK, Hancock J, Wennerstrom A, Haywood C, Meyers D, Johnson A, Polk M, Pesson CL, Seay JE, Stallard CN, Wells KB. A Rapid Assessment of Disaster Preparedness Needs and Resources during the COVID-19 Pandemic. Int J Environ Res Public Health. 2021 Jan 7;18(2):425. doi: 10.3390/ijerph18020425. PMID 33430355
- [Result] Everett A, Sugarman O, Wennerstrom A, et al. Community-informed strategies to address trauma and enhance resilience in climate-affected communities. Traumatology. 2020;26(3):285-297. doi:10.1037/trm0000225
- [Result] Pollock MJ, Wennerstrom A, True G, Everett A, Sugarman O, Haywood C, Johnson A, Meyers D, Sato J, Wells KB, Arevian AC, Massimi M, Berry J, Riefberg L, Onyewuenyi N, Springgate B. Preparedness and Community Resilience in Disaster-Prone Areas: Cross-Sectoral Collaborations in South Louisiana, 2018. Am J Public Health. 2019 Sep;109(S4):S309-S315. doi: 10.2105/AJPH.2019.305152. PMID 31505147
- See also: The official webpage for the C-LEARN study. Includes intervention materials, additional academic publications, presentations, and more. — http://www.c-learn.org

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT03977844/Prot_SAP_001.pdf